CLINICAL TRIAL: NCT07239518
Title: A Prospective Evaluation of Early Acupuncture for Immediate Continence Enhancement After Prostatectomy
Acronym: PEACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bin Xu (Other)
Responsible Party: Sponsor-Investigator, Bin Xu, Researcher, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025ZDSYLL366-P01
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Electroacupuncture Group (Experimental): Participants receive real electroacupuncture at acupoints including Shenshu (BL23), Pangguangshu (BL28), and Baliao (BL31-BL34). Treatment is administered for 30 minutes per session. It uses a continuous wave (starting at 2Hz) with a current intensity of 1-5mA, gradually increased to the maximum tolerable level for the patient.
  Interventions: Device: Electroacupuncture
- Sham Electroacupuncture (Sham Comparator): Participants receive sham acupuncture using non-penetrating, blunt-tipped placebo needles. These needles are applied at non-acupoint locations (1-2 cm away from real acupoints). Electrodes are attached to the sham needle handles, and the device is turned on (making noise/lighting up) but does not deliver any electrical current, to maintain blinding.
  Interventions: Device: Sham Electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture — Participants receive real electroacupuncture at acupoints including Shenshu (BL23), Pangguangshu (BL28), and Baliao (BL31-BL34). Treatment is administered for 30 minutes per session, for a total of 3 sessions (on post-operative days 7, 9, and 11). It uses a continuous wave (starting at 2Hz) with a current intensity of 1-5mA, gradually increased to the maximum tolerable level for the patient.
  Arms: Experimental: Electroacupuncture Group
Device: Sham Electroacupuncture — Participants receive sham acupuncture using non-penetrating, blunt-tipped placebo needles (e.g., Park or Streitberger needles). These needles touch the skin but do not penetrate. They are applied at non-acupoint locations (1-2 cm away from real acupoints) for 30 minutes per session, for a total of 3 sessions (on post-operative days 7, 9, and 11). Electrodes are attached to the sham needle handles, and the device is turned on (making noise/lighting up) but does not deliver any electrical current, to maintain blinding.
  Arms: Sham Electroacupuncture

SUMMARY:
This study is being done to see if early acupuncture treatment can help men control their urination better right after their urinary catheter is removed following prostate cancer surgery (radical prostatectomy).

Leaking urine is a very common problem immediately after this surgery, and current treatments often start after the catheter is already out. The researchers in this study believe that starting acupuncture before the catheter is removed might help "pre-activate" the nerves and muscles that control urination.

This is a prospective, multi-center, randomized, placebo-controlled study. The study plans to enroll 144 men who have had prostate cancer surgery. Participants will be randomly assigned (like flipping a coin) into two groups:

Treatment Group (72 participants): Will receive 3 sessions of real electroacupuncture.

Control Group (72 participants): Will receive 3 sessions of sham (placebo/fake) acupuncture. This involves using a special blunt needle that touches the skin but does not go in, and a machine that looks like it is on but provides no electricity.

The acupuncture or sham treatment will be given 3 times (on post-operative days 7, 9, and 11). The urinary catheter will be removed for all patients on post-operative day 14. All participants will also receive standard education on pelvic floor muscle exercises.

The main thing the researchers will measure (the primary endpoint) is the amount of urine leakage (in grams) during a 1-hour pad test, which will be done within the first week after the catheter is removed. Researchers will also check urinary control using questionnaires and other pad tests at 4, 8, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone radical prostatectomy with a confirmed pathological diagnosis of prostate cancer.
2. One week post-radical prostatectomy (RP).
3. Karnofsky Performance Score (KPS) ≥ 60 or ECOG Performance Status 0-1.
4. Age between 50 and 85 years.
5. Signed informed consent.

Exclusion Criteria:

1. Pathological results show positive surgical margins.
2. Previous treatment for post-operative urinary incontinence, such as cystostomy, urethral sphincter reconstruction, or urethral suspension.
3. Currently or within the last 6 months receiving treatment with principles similar to acupuncture (e.g., electroacupuncture, moxibustion, warm moxibustion).
4. Active urinary system infection (excluding asymptomatic lower urinary tract infection).
5. Known severe heart diseases, such as severe arrhythmia, severe heart failure, acute myocarditis, constrictive pericarditis, pericardial tamponade, severe valvular disease, or heart failure.
6. Known liver damage or potential severe liver disease (ALT or AST > 10 times the normal limit).
7. Known severe renal impairment (eGFR < 25mL/min/1.73m2), planned or ongoing dialysis, or acute contrast-induced nephropathy at screening.
8. Known dysfunction of other vital organs or severe primary diseases, such as hematopoietic system diseases.
9. Known coagulation dysfunction (with typical clinical diagnosis or clear laboratory test results).
10. Patients with mental illness or cognitive impairment; patients with severe depression, alcohol dependence, or a history of drug abuse.
11. Urinary incontinence known to be due to other reasons.
12. According to the investigator's judgment, the patient is not suitable for this study or has a high probability of dropout (e.g., frequent changes in work environment that make follow-up difficult).
13. Life expectancy ≤ 6 months, as judged by the investigator.
14. Currently participating in other clinical trials.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Urine Leakage Amount from 1-Hour Pad Test | At the 1-week follow-up visit after catheter removal.
  Urine leakage volume, measured in grams (g), collected during a standardized 1-hour pad test.

SECONDARY OUTCOMES:
1-Hour Pad Test Urine Leakage Amount (Later Follow-ups) | At 4-week and 24-week follow-up visits after catheter removal.
ICIQ-SF (International Consultation on Incontinence Questionnaire - Short Form) Score | At 1, 4, 8, 12, and 24-week follow-up visits after catheter removal.
Proportion of Completely Continent (Leak-Free) Patients | At 1, 4, 8, 12, and 24-week follow-up visits after catheter removal.
SAS (Self-Rating Anxiety Scale) Score | At 1, 4, 8, 12, and 24-week follow-up visits.
IPSS (International Prostate Symptom Score), based on voiding diaries | At 1, 4, 8, 12, and 24-week follow-up visits.

DOCUMENTS (2):
  • Study Protocol (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT07239518/Prot_000.pdf
  • Informed Consent Form (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT07239518/ICF_001.pdf